CLINICAL TRIAL: NCT05177757
Title: Feasibility of a Yoga Program for Veterans With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marquette University (Other)
Responsible Party: Principal Investigator, Jacklynn Fitzgerald, Assistant Professor, Marquette University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR- 3973
Record Dates: First submitted 2021-11-10; First posted 2022-01-05 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga Intervention (Experimental): The yoga exercise program will be conducted at the Marquette campus and will consist of one session per week for 12 weeks. The duration of each session will be approximately one hour. The program the investigators will use is the Mindful Resilience for Trauma Recovery Program (https://www.veteransyogaproject.org/), an evidence-informed practice adapted for veterans with PTSD based on clinical and neuroscientific knowledge. This program is a 12-week protocol developed by a licensed clinical psychologist and is publicly available. All yoga sessions will be standardized based on the resilience program guidelines.
  Interventions: Other: Yoga Intervention

INTERVENTIONS:
Other: Yoga Intervention — The yoga exercise program will be conducted at the Marquette campus and will consist of one session per week for 12 weeks. The duration of each session will be approximately one hour. The program the investigators will use is the Mindful Resilience for Trauma Recovery Program (https://www.veteransyogaproject.org/), an evidence-informed practice adapted for veterans with PTSD based on clinical and neuroscientific knowledge. This program is a 12-week protocol developed by a licensed clinical psychologist and is publicly available. All yoga sessions will be standardized based on the resilience program guidelines.

SUMMARY:
This study is designed to examine the feasibility of a 12-week yoga program on physiological and psychological health and its neurobiological mechanisms in N=15 veterans with posttraumatic stress disorder (PTSD). The investigators will be examining specific parameters of health and mechanisms before and after the yoga program.

ELIGIBILITY:
Inclusion Criteria:

* U.S. Military Veteran
* 18 years of age or older
* Diagnosis of PTSD as assessed by a score of >30 on the PTSD-Checklist Version 5 (PCL-5)
* Willing and able to attend testing and yoga sessions at the Athletic and Human Research Performance Center (AHPRC) on the campus of Marquette University
* Clear to participate in physical activity based on the Physical Activity Readiness Questionnaire (PARQ+)

Exclusion Criteria:

* Currently pregnant or trying to become pregnant
* Positive score to one or more items on the PAR-Q+ without physician approval
* Already established regular use of yoga (i.e., more than one day per week)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-28 (Actual)

PRIMARY OUTCOMES:
Endocannabinoid assay | Change in ligands from baseline to12 weeks
  Endocannabinoid ligands reported in ng/ml
Cortisol assay | Change in cortisol from baseline to12 weeks
  Cortisol reported in μg/dL
Cognitive functioning using a computerized battery | Change in performance from baseline to12 weeks
  Performance on cognitive tasks reported in accuracy and reaction time
Body Mass Index (BMI) | Change in BMI from baseline to12 weeks
  Body Mass Index (BMI) calculated by height and weight
Blood pressure | Change in blood pressure from baseline to12 weeks
  Blood pressure reported in systolic and diastolic (mmHg)
Heart rate | Change in heart rate from baseline to12 weeks
  Heart rate reported in beats per minute (BPM)
Heart rate variability (HRV) | Change in HRV from baseline to12 weeks
  Heart rate variability (HRV) reported in the standard deviation of the RR intervals (distance between heartbeats) as quantified on standard electrocardiogram (ECG)
Lung functioning | Change in lung functioning from baseline to12 weeks
  Lung functioning measured by spirometry reported in vital capacity (VC)
Range of motion | Change in range of motion from baseline to12 weeks
  Range of motion measured by goniometer reported in degrees
Body composition | Change in body composition from baseline to12 weeks
  Body composition measured by dual-energy x-ray absorptiometry (DEXA) reported in volume cubic meters (m3) and mass (kilograms)
Hand grip strength | Change in hand grip strength from baseline to12 weeks
  Hand grip strength measured by a dynamometer reported in pounds (lbs)
Aerobic fitness | Change in aerobic fitness from baseline to12 weeks
  Aerobic fitness measured by a submaximal graded exercise test reported in the volume of oxygen consumed (VO2)
Physical activity | Change in physical activity from baseline to12 weeks
  Physical activity measured by a accelerometer reported in change in velocity over time (meters per seconds)
Severity of posttraumatic stress disorder (PTSD) | Change in scores from baseline to12 weeks
  Scores on the Clinician Administered PTSD Scale (CAPS-5) (range 0-80; higher scores indicate more severity)
Frequency of physical activity | Change in scores from baseline to12 weeks
  Scores on the International Physical Activity Questionnaire-Short Form (IPAQ-SF) reported in hours and minutes each day
Physical health rating | Change in scores from baseline to12 weeks
  Scores on the Medical Outcomes Study-Short Form (SF-36) (range 0-100; higher scores indicate better health outcome)
Severity of sleep disturbance | Change in scores from baseline to12 weeks
  Scores on the Pittsburgh Sleep Quality Index (PSQI) (range 0-21; higher scores indicate worse sleep quality)
Mindfulness rating | Change in scores from baseline to12 weeks
  Scores on the Five Facet Mindfulness Questionnaire (FFMQ) (range 39-195; higher scores indicate more mindfulness)
Frequency of yoga rating | Change in scores from baseline to12 weeks
  Scores on the Yoga and Self-efficacy Scale (YSES) (range 12-108; higher scores indicate more engagement with yoga practices)

CONTACTS AND LOCATIONS:
Overall Officials: Jacklynn Fitzgerald, PhD, Principal Investigator — Marquette University
Locations (1):
- Marquette University, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No